CLINICAL TRIAL: NCT04057092
Title: Perioperative Immunonutrition in Patients Undergoing Gynecologic or General Elective Surgery (PURPOSE): a Feasibility Trial
Brief Title: Perioperative Immunonutrition in Patients Undergoing Gynecologic or General Elective Surgery (PURPOSE)
Acronym: PURPOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Principal Investigator, Limor Helpman, Associate Professor, Hamilton Health Sciences Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-4462
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Surgical Site Infection; Post-Op Complication
Keywords: perioperative immunonutrition; clinical nutrition; infection prevention
MeSH Terms: conditions — Surgical Wound Infection; Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Eligible and consenting gynecologic oncology and general surgery patients will receive EMN's nutritional supplement INergy-FLD® both before and after elective surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Eligible patients undergoing gynecologic oncology or general surgery will receive perioperative immunonutrition supplement INergy-FLD®. The operation should occur within 8 weeks from enrolment in the pilot study. Upon assessment and enrolment in the pilot study, patients will have a consultation with their physician in the preoperative clinic and will be provided with 10 days worth of INergy-FLD® beverages, 30 servings total.
  Interventions: Dietary Supplement: Dietary Supplement INergy-FLD

INTERVENTIONS:
Dietary Supplement: Dietary Supplement INergy-FLD — INergy-FLD® is an immune modulating formula containing various ingredients including L-Arginine, whey protein isolate, and omega-6 fatty acid, aimed to attenuate excessive inflammatory responses without being immunosuppressive and to replenish nutrients that are depleted in a state of surgical stress, thereby enhancing the recovery process and decreasing the risk of infection. The volume of the beverage is 250mL per serving and patients will be asked to consume 3 servings periodically per day for 5 days prior to surgery and 5 days following surgery.
  Other Names: INergy-FLD®

SUMMARY:
The objective of the implementation pilot is to assess the practicality of introducing a perioperative immunonutrition protocol into a hospital environment as well as a true measure of impact on the rate of surgical site infection (SSI).

DETAILED DESCRIPTION:
Postoperative infectious complications are independently associated with increased hospital length of stay (LOS) and cost, and contribute to significant inpatient morbidity. Despite recent advances in surgical techniques and perioperative management, the rate of postoperative infectious complications remains high with 54% of all hospital-acquired-infections occurring in high-risk surgical populations.2 Poor nutritional status along with surgical stress predisposes patients to postoperative complications and immune depression. Research is now demonstrating the importance of additional perioperative nutritional support through the use of enteral and parenteral feeds in high-risk patients, with a specific focus on the role of immunonutrition. Immunonutrition substrates have been found to modulate postsurgical immuno-depression and inflammatory responses and positively impact patient outcomes.

Immunonutrition is defined as a solution that contains nutrients such as arginine, omega fatty acids, and protein. Arginine deficiency after surgical stress was first reported over 30 years ago, and recent studies have demonstrated that the perioperative use of arginine-supplemented diets have the ability to decrease the rate of postoperative infection. Arginine is an amino acid that is synthesized in the body but not in high enough concentration to support metabolic needs during periods of stress, such as surgery. While under stress, arginine is the primary fuel source for T-cells and helps maintain immune function and decrease the risk of infection. Th1 induced macrophages also use arginine for many of their immune functions. In addition, omega fatty acids, such as n-6 and n-3, are derived from fish oil and have been shown to attenuate the production of inflammatory compounds and ultimately reduce the cytotoxicity of inflammatory cells. This role that omega fatty acids play in the resolution of inflammation results in enhanced wound healing and improved lymphocyte function. Finally, whey protein substrates have great potential to be used effectively to support post-surgery anabolism. Whey proteins are of high quality, have proved to be effective in modulating muscle protein synthesis, and are a convenient way to supplement protein needs in malnourished patients. Whey proteins also have immuno-modulating properties, including biosynthesis of antioxidant glutathione, which could attenuate the catabolic effects of surgery and spare protein. These ingredients have been shown to work synergistically and are associated with significantly better overall and recurrence-free survival. Each element works towards improving the immune response through modulation of excessive inflammatory responses and replenishing depleted nutrients when the body is in a state of surgical stress.13

The HHS implementation pilot will provide preoperative patients with EMN's immunonutrition formula, INergy-FLD®. INergy-FLD® is an immune-modulating solution that contains whey protein isolate, refined fish oil with omega 6 fatty acids, antioxidants such as vitamins A, C, D and E, and has an elevated amino acid concentration with 4.2 grams of L-Arginine per serving. It has a natural citrus flavor, low sugar and a trace of lactose, and therefore can be tolerated by patients who are lactose intolerant. INergy-FLD® is categorized under Health Canada as a formulated liquid diet (FLD). INergy-FLD® complies with the detailed and explicit compositional and labeling requirements of an FLD supplement as well as providing complete directions for preparation and the use of the food product (Food Category: CFIA)

Patient reported consumption diaries will be used to track the consumption of INergy-FLD® by patients in the perioperative period, and patient feedback will be sought on experience and barriers in implementation of this regimen. In order to track the impact of INergy-FLD® on the rate of postoperative infectious complications, HHS will rely on the NSQIP patient-outcome audit system. According to two new studies presented by researchers from the American College of Surgeons (ACS), NSQIP provides more accurate data than administrative data for driving surgical quality improvement. NSQIP codes are standardized, very specific, and can identify the primary reason for readmission. Other advantages of NSQIP include the detail of preoperative risk variables collected by the database, allowing for a more robust risk-adjusted analysis. Using this database available at HHS, EMN will be able to accurately analyze the impact of INergy-FLD® immunonutrition on surgical patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 years of age or older who are undergoing gynecologic oncology or general surgery (including resectable types of cancer) for which an elective operation is planned.
* Patients who are lactose intolerant are eligible for the study because the amount of lactose in INergy-FLD® is minimal (trace).

Exclusion Criteria:

* Cannot tolerate enteral intake
* Organ failure (liver, kidney)
* Patients currently on steroids
* Female patients who are pregnant and/or lactating
* Galactosemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of compliance to protocol | 5 days postoperative
  a visual assessment of empty nutrition packages, to ensure patient has consumed 70% or more of the nutrition supplements

SECONDARY OUTCOMES:
Surgery site infection (SSI) | 30 days postoperative
  SSI's will be determined and tracked by NSQIP following the patients' hospital stay and up to 30 days from the initial operation including superficial, fascia, and deep infections. The NSQIP is not a measure, but rather a program by which hospitals report surgical outcomes including infections. The outcome of importance will be the number of surgery site infections reported by each group
Length of hospital stay | up to 12 weeks.
  Number of days hospital stay post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Juravinski Cancer Centre, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No